CLINICAL TRIAL: NCT02481024
Title: 'Moving From Hospital to Home' - Exploring the Impact of Care Transition on Medication Adherence in Cardiac Patients: a Qualitative Study Protocol
Brief Title: Impact of Care Transition on Medication Adherence in Cardiac Patients
Status: Completed | Type: Observational
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: V1_18_06_15
Record Dates: First submitted 2015-06-18; First posted 2015-06-25 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2016-08

CONDITIONS: Acute Coronary Syndrome
Keywords: Qualitative; Care transition; Medication
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Background:

Medication adherence following acute coronary syndrome (ACS) is often sub-optimal. Poor adherence is associated with increased risk of rehospitalisation along with higher rates of morbidity and mortality. After a cardiac event, transitioning from hospital into primary care can be problematic if it is not organised or coordinated properly. Patients can often find themselves unprepared and lacking the necessary information for self-management of their disease. The impact of care transition on medication adherence has not been studied in ACS.

Objectives:

This study will explore how an ACS patients' journey from hospital into primary care affects medicines use. Further, to understand how medicine information is communicated and how this influences patient beliefs about medicines.

Methods:

This is an interview study with recently hospitalised ACS patients discussing medication beliefs, communication of medicine information and the challenges when transitioning from specialist to primary care. Patients will be recruited from Guy's and St Thomas' NHS Foundation Trust and telephone interviews will be scheduled 3-4 weeks post-discharge. An inductive thematic analysis will be used to identify, construct and analyse patterns in the data and to develop a framework analysis. Analysis will be an iterative process conducted in parallel with data collection to highlight when data saturation has been reached.

Dissemination:

The primary objective is to develop a pharmacist-led behaviour change intervention to improve rates of medication adherence following an ACS. The in-depth patient data collected in this current study will contribute to the design and development of the intervention. Understanding the research topic from the patients' perspective is a necessity when designing an intervention targeting behaviour change.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age
* have a confirmed index diagnosis of ACS
* have sufficient spoken English to partake in an interview

Exclusion Criteria:

* under 18 years of age
* lack the level of spoken English required to be interviewed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalised after an acute coronary syndrome event.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2015-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Patient experiences | 3-4 weeks after discharged from hospital
  Analysing patients' experiences of care transition and its impact on adherence and treatment beliefs. This will be done using thematic analysis to identify, construct and assess patterns in the qualitative data to develop a framework analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom